CLINICAL TRIAL: NCT00195208
Title: A Randomized, 2-Period, Crossover, Pharmacodynamic Comparability Study Comparing A Pantoprazole Spheroid Formulation to the Currently Marketed Tablet Formulation in Subjects With GERD and a History of Erosive Esophagitis.
Brief Title: Study Comparing a Pantoprazole Formulation to the Currently Marketed Tablet for GERD and Erosive Esophagitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 3001B1-332
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Gastroesophageal Reflux; Esophagitis
Keywords: Gastroesophageal Reflux Disease (GERD)
MeSH Terms: conditions — Gastroesophageal Reflux; Esophagitis | interventions — Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole for approximately 9 weeks

SUMMARY:
The purpose of this study is to demonstrate pharmacodynamic comparability between the pantoprazole spheroid formulation and the marketed tablet formulation.

ELIGIBILITY:
Inclusion Criteria:

* GERD and a history of Erosive Esophagitis documented by endoscopy
* H. pylori negative

Exclusion Criteria:

* Gastrointestinal conditions such as esophageal stricture, esophageal varices, previous vagotomy
* Achlorhydria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2005-06; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Comparison of MAO between the two formulations.

SECONDARY OUTCOMES:
Comparison of BAO and pH parameters between the two formulations.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (7):
- United States (7):
  - Anaheim, California
  - Los Angeles, California
  - Orange, California
  - San Diego, California
  - Miami, Florida
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania